CLINICAL TRIAL: NCT02497144
Title: Effects of Neuromuscular Electrical Stimulation on Functional Exercise Capacity and Quality of Life in Patients With Interstitial Lung Disease
Brief Title: Neuromuscular Electrical Stimulation in Patients With Interstitial Lung Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Assoc. Prof, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Gazi University3
Record Dates: First submitted 2015-07-08; First posted 2015-07-14 (Estimated); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Interstitial Lung Disease
Keywords: interstitial lung disease; neuromuscular electrical stimulation; exercise capacity; quality of life
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NMES Group (Active Comparator): Intervention: NMES group will receive neuromuscular electrical stimulation using high frequency galvanic stimulation and breathing exercises.
  Neuromuscular electrical stimulation will be applied bilaterally to quadriceps femoris muscle for 3days/6 weeks by a physiotherapist.
  NMES group will also perform breathing exercises 120 times/day, 7 days/week, for 6 weeks.
  Interventions: Other: NMES Group
- Control Group (Sham Comparator): Sham: Control group will receive breathing exercises. Control group will perform breathing exercises 120 times/day, 7 days/week, for 6 weeks.
  Control group will be followed-up by telephone once a week.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: NMES Group — Neuromuscular electrical stimulation
  Arms: NMES Group
Other: Control Group — Breathing exercises
  Arms: Control Group

SUMMARY:
Decreased exercise capacity and quality of life, increased dyspnea and fatigue perception and hypoxemia during exercise is seen in patients with interstitial lung disease. Impaired ventilatory response, increased lung compliance, ventilation-perfusion mismatching and inadequate peripheral circulation causes decreased exercise capacity. Another important factor that induce decreased exercise capacity is peripheral muscle weakness. In literature, there is no study investigated effects of neuromuscular electrical stimulation on functional exercise capacity, respiratory and peripheral muscle strength, pulmonary functions, physical activity level, dyspnea and fatigue perception in patients with interstitial lung disease.

DETAILED DESCRIPTION:
In literature, there was increased quantity of study investigated effects of neuromuscular electrical stimulation in chronic lung disease patients. It was used as a pulmonary rehabilitation component especially in patients with decreased exercise capacity and peripheral muscle strength, intensely increased dyspnea inhibits exercise. It was demonstrated that neuromuscular electrical stimulation improved functional exercise capacity, peripheral muscle strength and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with interstitial lung disease
* Clinically stable
* Under standard medication
* Having no exacerbation or infection

Exclusion Criteria:

* Cognitive disorders
* Orthopedic and neurological problems
* Contraindications to apply the neuromuscular electrical stimulation (pace maker, sensory defects, etc...)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-07-15; Primary Completion 2018-09-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Functional exercise capacity | 6 weeks
  Six minute walk test

SECONDARY OUTCOMES:
Pulmonary functions | 6 weeks
  Spirometry
Inspiratory and expiratory muscle strength (MIP,MEP) | 6 weeks
  Mouth pressure device
Dyspnea | 6 weeks
  Modified Borg and Modified Medical Research Council (MMRC) Dyspnea scales
Peripheral muscle strength | 6 weeks
  Hand held dynamometer
Maximal exercise capacity | 6 weeks
  Incremental shuttle walk test
Fatigue | 6 weeks
  Fatigue Severity Scale
Physical activity | 6 weeks
  Metabolic holter
Cough related quality of life | 6 weeks
  Leicester Cough Questionnaire
Depression | 6 weeks
  Montgomery Asberg Depression Rating Scale (MADRS) (Turkish versions of all scales)
Generic quality of life | 6 weeks
  Short Form (SF-36) Health Survey
Disease specific quality of life | 6 weeks
  Saint George Quality of Life Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Meral Boşnak-Güçlü, PhD, Study Chair — Gazi University; Burcu Camcıoğlu, MSc, Study Director — Gazi University; Müşerrefe N Karadallı, MSc, Principal Investigator — Gazi University; Deran Oskay, PhD, Principal Investigator — Gazi University; Haluk Türktaş, Dr, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

REFERENCES:
- [Result] Swigris JJ, Gould MK, Wilson SR. Health-related quality of life among patients with idiopathic pulmonary fibrosis. Chest. 2005 Jan;127(1):284-94. doi: 10.1378/chest.127.1.284. PMID 15653996
- [Result] Lama VN, Flaherty KR, Toews GB, Colby TV, Travis WD, Long Q, Murray S, Kazerooni EA, Gross BH, Lynch JP 3rd, Martinez FJ. Prognostic value of desaturation during a 6-minute walk test in idiopathic interstitial pneumonia. Am J Respir Crit Care Med. 2003 Nov 1;168(9):1084-90. doi: 10.1164/rccm.200302-219OC. Epub 2003 Aug 13. PMID 12917227
- [Result] Spruit MA, Thomeer MJ, Gosselink R, Troosters T, Kasran A, Debrock AJ, Demedts MG, Decramer M. Skeletal muscle weakness in patients with sarcoidosis and its relationship with exercise intolerance and reduced health status. Thorax. 2005 Jan;60(1):32-8. doi: 10.1136/thx.2004.022244. PMID 15618580
- [Result] Vivodtzev I, Lacasse Y, Maltais F. Neuromuscular electrical stimulation of the lower limbs in patients with chronic obstructive pulmonary disease. J Cardiopulm Rehabil Prev. 2008 Mar-Apr;28(2):79-91. doi: 10.1097/01.HCR.0000314201.02053.a3. PMID 18360183
- [Result] Bourjeily-Habr G, Rochester CL, Palermo F, Snyder P, Mohsenin V. Randomised controlled trial of transcutaneous electrical muscle stimulation of the lower extremities in patients with chronic obstructive pulmonary disease. Thorax. 2002 Dec;57(12):1045-9. doi: 10.1136/thorax.57.12.1045. PMID 12454299
- [Result] Sillen MJH, Speksnijder CM, Eterman RA, Janssen PP, Wagers SS, Wouters EFM, Uszko-Lencer NHMK, Spruit MA. Effects of neuromuscular electrical stimulation of muscles of ambulation in patients with chronic heart failure or COPD: a systematic review of the English-language literature. Chest. 2009 Jul;136(1):44-61. doi: 10.1378/chest.08-2481. Epub 2009 Apr 10. PMID 19363213